CLINICAL TRIAL: NCT04562467
Title: The Icosapent Ethyl and Prevention of Vascular Regenerative Cell Exhaustion Study
Brief Title: The Use of Icosapent Ethyl on Vascular Progenitor Cells in Individuals With Elevated Cardiovascular Risk
Acronym: IPE-PREVENTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: HLS Therapeutics, Inc (Unknown); Unity Health Toronto (Other); Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00043561
Record Dates: First submitted 2020-09-13; First posted 2020-09-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Triglycerides High; Diabetes Mellitus, Type 2
Keywords: Cardiometabolic Risk; Type 2 Diabetes; Icosapent Ethyl; Omega-3; Vascular Diseases; Progenitor Cells; Vascular Disease; Blood Lipids
MeSH Terms: conditions — Cardiovascular Diseases; Hypertriglyceridemia; Diabetes Mellitus, Type 2; Vascular Diseases | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Icosapent Ethyl + Standard of Care (Experimental): Icosapent Ethyl 1000 MG Oral Capsule [Vascepa] 2 x 1g capsules BID (4g total) as per REDUCE-IT
  Interventions: Drug: Icosapent Ethyl 1000 MG Oral Capsule [Vascepa]
- Standard of Care (No Intervention): Standard of care therapy (including statin therapy as per inclusion criteria)

INTERVENTIONS:
Drug: Icosapent Ethyl 1000 MG Oral Capsule [Vascepa] — 2 x 1g capsules BID as per REDUCE-IT
  Other Names: Vascepa; IPE
  Arms: Icosapent Ethyl + Standard of Care

SUMMARY:
IPE-PREVENTION is a prospective, randomized, 3-month long, open-label study. A total of 70 individuals with elevated cardio-metabolic risk and heightened triglyceride levels, and who are on stable statin therapy will be randomized (1:1) to receive either icosapent ethyl (IPE) 2g BID or standard of care.

It is hypothesized that assignment to IPE will lower progenitor cell depletion as well as limit progenitor cell dysfunction. This study may offer some molecular and cellular insights into the mechanisms underlying the cardiovascular benefits of IPE therapy reported in the REDUCE-IT trial.

DETAILED DESCRIPTION:
The development and natural history of atherothrombosis involves the pathophysiological interplay between inflammation, dyslipidemia, oxidative stress and endothelial dysfunction. Unregulated, these processes culminate in endothelial dysfunction, and ultimately cardio-metabolic chronic diseases. Aberrant lipid oxidation due to elevated triglycerides and cholesterol primes and activates innate immune cell activity resulting in elevated inflammation and oxidative stress.

The randomized, placebo-controlled REDUCE-IT trial enrolled individuals with established atherosclerotic heart disease, or diabetes and an additional risk factor, who were on pre-existing statin therapy with persistent hypertriglyceridemia. REDUCE-IT reported that the group allocated to the omega-3 fatty acid icosapent ethyl (IPE; 2g BID) exhibited a 25% relative risk reduction for the primary composite endpoint of CV death, nonfatal myocardial infarction, nonfatal stroke, coronary revascularization, or unstable angina, and a 20% decreased risk of CV death when compared to standard of care. Vascepa® (IPE) is currently approved by Health Canada and the U.S. FDA for the reduction of cardiovascular risk in statin-treated individuals with elevated triglycerides who are either at heightened cardiovascular risk or who have diabetes and at least one risk factor.

The exact mechanism through which IPE decreased cardiovascular events in REDUCE-IT has not yet been elucidated.

The population and function of circulating pro-vascular progenitor cells have been shown to benefit from diminished lipid oxidation, inflammation and oxidative stress. A healthy population of circulating pro-vascular progenitor cells in turn affords timely and efficient blood vessel repair, regeneration and atheroprotection.

The omega-3 fatty acid eicosapentaenoic acid (EPA) has been reported to inhibit M1 macrophage polarization in a murine model and increase human endothelial progenitor cell (EPC) colony formation and functionality in vitro. In vivo, EPA levels have been observed to correlate significantly with circulating EPC number (CD34+CD133+VEGFR2+ cells). Collectively, these findings affirm that EPA, and potentially omega-3 fatty acids, can enhance the number and function of circulating pro-vascular progenitor cells and can alter M1/M2 macrophage balance towards a regenerative blood vessel phenotype.

IPE-PREVENTION is a prospective, 3-month long, open-label study that will randomize a total of 70 individuals with elevated cardio-metabolic risk and heightened triglyceride levels and who are on stable statin therapy to either IPE 2g BID or standard of care. Blood samples will be collected at the baseline and month 3 visits for evaluations of cell populations in the blood as well as measurements of biomarkers that contribute to the proinflammatory and pro-oxidant milieu of individuals at elevated cardio-metabolic risk. The study will utilize the AldefluorTM assay to differentiate between and enumerate hematopoietic progenitor cells, EPCs, granulocyte precursors and macrophage precursors. The overarching goal would be to document how assignment to IPE and standard-of-care impact on circulating progenitor cell depletion and dysfunction. The effect of IPE exposure on the inflammatory and oxidative profile will also be assessed.

The results of this investigation may offer some molecular and cellular insights into the mechanisms underlying the cardiovascular benefits of IPE therapy reported in the REDUCE-IT trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥65 years of age and men ≥40 years of age with established CVD (see criterion 'a' below) or ≥50 years of age with diabetes and one additional CV risk factor (see criterion 'b' below)

   1. Those with established CVD should have ≥1 of the following clinical history

      * Documented coronary artery disease (CAD)

        * Prior MI
        * Multivessel CAD (≥50% stenosis in ≥2 major epicardial coronary arteries)
        * Hospitalization for high-risk non-ST-segment elevation acute coronary syndrome
      * Documented cerebrovascular or carotid disease (≥1 of the following)

        * Prior ischemic stroke
        * Carotid artery disease with ≥50% stenosis
        * History of carotid revascularization
      * Documented peripheral artery disease (≥1 of the following)

        * Ankle-brachial index (ABI) <0.9 with symptoms of intermittent claudication
        * History of aorto-iliac or peripheral arterial intervention
   2. Those with a history of diabetes (either type 1 or type 2 diabetes mellitus) but no CVD should also have ≥1 of the following:

      * Cigarette smoker or stopped smoking within 3 months before the baseline visit
      * Documented hypertension OR on antihypertensive agents
      * HDL-C ≤1.0 mmol/L for men or ≤1.3 mmol/L for women
      * High sensitivity C-reactive protein >3.0 mg/L
      * eGFR 30 to 60 mL/min/1.73m2
      * Documented micro- or macro-albuminuria
      * Retinopathy

        * Non-proliferative retinopathy
        * Preproliferative or proliferative retinopathy
        * Maculopathy
        * Advanced diabetic retinopathy
        * History of photocoagulation
      * ABI <0.9 without symptoms of intermittent claudication
2. Elevated triglycerides (≥1.5 mmol/L but <5.6 mmol/L)
3. On stable statin therapy for ≥4 weeks at the baseline visit
4. Willing to provide written informed consent and be compliant with the study requirements
5. Willing and able to follow the diet recommended by the study doctor

Exclusion Criteria:

1. Participation in another clinical trial with an investigational agent ≤90 days prior to screening
2. Women who are of childbearing potential
3. Any condition or therapy which the study doctor thinks might pose a risk to the participant
4. Severe (New York Heart Association class IV) heart failure
5. Any life-threatening disease expected to result in death within the next 2 years
6. Diagnosis or laboratory evidence of active severe liver disease
7. HbA1c >10.0% at the baseline visit
8. SBP ≥200 mmHg or DBP ≥100 mmHg (despite being on antihypertensive therapy)
9. Planned coronary intervention or any non-cardiac major surgical procedure
10. Known familial lipoprotein lipase deficiency, apolipoprotein C-II deficiency, or familial dysbetalipoproteinemia
11. Statin intolerant or hypersensitivity to statin therapy
12. Require peritoneal dialysis or hemodialysis
13. eGFR <30 mL/min/1.73m2
14. History of atrial fibrillation
15. History of major bleeding event(s)
16. Documented history of pancreatitis
17. Malabsorption syndrome and/or chronic diarrhea
18. Known acquired immunodeficiency syndrome
19. Unexplained elevated creatine kinase concentration >5 × the upper limits of normal or elevation due to known muscle disease
20. Use of niacin, fibrates, omega-3 fatty acids, dietary supplements containing omega-3 fatty acids, bile acid sequestrants or PCSK9 inhibitors
21. Known hypersensitivity to fish and/or shellfish, or ingredients of IPE
22. Inability to swallow IPE capsules whole
23. Drug or alcohol abuse within the past 6 months, and inability/unwillingness to abstain from drug abuse and excessive alcohol consumption during the study
24. Mental/psychological concerns or any other reason to expect difficulty in complying with the study requirements or understanding the goal and potential risks of being a part of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of ALDHhiSSClowCD133+ cells in individuals treated with IPE compared to SOC for 3 months | Baseline - 3 months post-randomization

OTHER OUTCOMES:
Change in the ratio of ALDHhiSSCmid pro-inflammatory:anti-inflammatory monocyte precursor cells in individuals treated with IPE compared to SOC for 3-months. | Baseline - 3 months post-randomization
Change in the mean frequency of ALDHhiSSChi cells in individuals treated with IPE compared to SOC for 3-months. | Baseline - 3 months post-randomization
Changes in the concentration of serum oxidative stress markers from baseline to the 3-month visit in individuals treated with IPE compared to SOC | Baseline - 3 months post-randomization
Changes in the concentration of serum inflammatory markers from baseline to the 3-month visit in individuals treated with IPE compared to SOC | Baseline - 3 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — Unity Health Toronto; David A Hess, PhD, Principal Investigator — Robarts Research Institute, London, Ontario; Deepak L Bhatt, MD, MPH, Study Chair — Brigham and Women's Hospital, Boston, Massachusetts
Locations (3):
- Canada (3):
  - The Oshawa Clinic, Oshawa, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario
  - Langstaff Medical Clinic, Vaughan, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mechanick JI, Farkouh ME, Newman JD, Garvey WT. Cardiometabolic-Based Chronic Disease, Adiposity and Dysglycemia Drivers: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Feb 11;75(5):525-538. doi: 10.1016/j.jacc.2019.11.044. PMID 32029136
- [Background] Carmeliet P. Angiogenesis in health and disease. Nat Med. 2003 Jun;9(6):653-60. doi: 10.1038/nm0603-653. PMID 12778163
- [Background] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Cardiovascular Risk Reduction with Icosapent Ethyl for Hypertriglyceridemia. N Engl J Med. 2019 Jan 3;380(1):11-22. doi: 10.1056/NEJMoa1812792. Epub 2018 Nov 10. PMID 30415628
- [Background] Isner JM, Asahara T. Angiogenesis and vasculogenesis as therapeutic strategies for postnatal neovascularization. J Clin Invest. 1999 May;103(9):1231-6. doi: 10.1172/JCI6889. No abstract available. PMID 10225965
- [Background] Peichev M, Naiyer AJ, Pereira D, Zhu Z, Lane WJ, Williams M, Oz MC, Hicklin DJ, Witte L, Moore MA, Rafii S. Expression of VEGFR-2 and AC133 by circulating human CD34(+) cells identifies a population of functional endothelial precursors. Blood. 2000 Feb 1;95(3):952-8. PMID 10648408
- [Background] Takamura M, Kurokawa K, Ootsuji H, Inoue O, Okada H, Nomura A, Kaneko S, Usui S. Long-Term Administration of Eicosapentaenoic Acid Improves Post-Myocardial Infarction Cardiac Remodeling in Mice by Regulating Macrophage Polarization. J Am Heart Assoc. 2017 Feb 21;6(2):e004560. doi: 10.1161/JAHA.116.004560. PMID 28223437
- [Background] Devaraj S, Chien A, Rao B, Chen X, Jialal I. Modulation of endothelial progenitor cell number and function with n-3 polyunsaturated fatty acids. Atherosclerosis. 2013 May;228(1):94-7. doi: 10.1016/j.atherosclerosis.2013.02.036. Epub 2013 Mar 13. PMID 23528830
- [Background] Morishita T, Uzui H, Ikeda H, Amaya N, Kaseno K, Ishida K, Fukuoka Y, Lee JD, Tada H. Association of CD34/CD133/VEGFR2-Positive Cell Numbers with Eicosapentaenoic Acid and Postprandial Hyperglycemia in Patients with Coronary Artery Disease. Int J Cardiol. 2016 Oct 15;221:1039-42. doi: 10.1016/j.ijcard.2016.07.079. Epub 2016 Jul 5. PMID 27447811
- [Background] Capoccia BJ, Robson DL, Levac KD, Maxwell DJ, Hohm SA, Neelamkavil MJ, Bell GI, Xenocostas A, Link DC, Piwnica-Worms D, Nolta JA, Hess DA. Revascularization of ischemic limbs after transplantation of human bone marrow cells with high aldehyde dehydrogenase activity. Blood. 2009 May 21;113(21):5340-51. doi: 10.1182/blood-2008-04-154567. Epub 2009 Mar 26. PMID 19324906
- [Background] Putman DM, Liu KY, Broughton HC, Bell GI, Hess DA. Umbilical cord blood-derived aldehyde dehydrogenase-expressing progenitor cells promote recovery from acute ischemic injury. Stem Cells. 2012 Oct;30(10):2248-60. doi: 10.1002/stem.1206. PMID 22899443
- [Background] Terenzi DC, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Circulating Pro-Vascular Progenitor Cell Depletion During Type 2 Diabetes: Translational Insights Into the Prevention of Ischemic Complications in Diabetes. JACC Basic Transl Sci. 2018 Nov 5;4(1):98-112. doi: 10.1016/j.jacbts.2018.10.005. eCollection 2019 Feb. PMID 30847424
- [Background] Hess DA, Terenzi DC, Trac JZ, Quan A, Mason T, Al-Omran M, Bhatt DL, Dhingra N, Rotstein OD, Leiter LA, Zinman B, Sabongui S, Yan AT, Teoh H, Mazer CD, Connelly KA, Verma S. SGLT2 Inhibition with Empagliflozin Increases Circulating Provascular Progenitor Cells in People with Type 2 Diabetes Mellitus. Cell Metab. 2019 Oct 1;30(4):609-613. doi: 10.1016/j.cmet.2019.08.015. Epub 2019 Aug 30. PMID 31477497
- [Background] Balber AE. Concise review: aldehyde dehydrogenase bright stem and progenitor cell populations from normal tissues: characteristics, activities, and emerging uses in regenerative medicine. Stem Cells. 2011 Apr;29(4):570-5. doi: 10.1002/stem.613. PMID 21308868
- [Background] Gentry T, Foster S, Winstead L, Deibert E, Fiordalisi M, Balber A. Simultaneous isolation of human BM hematopoietic, endothelial and mesenchymal progenitor cells by flow sorting based on aldehyde dehydrogenase activity: implications for cell therapy. Cytotherapy. 2007;9(3):259-74. doi: 10.1080/14653240701218516. PMID 17464758
- [Background] Shoulars K, Noldner P, Troy JD, Cheatham L, Parrish A, Page K, Gentry T, Balber AE, Kurtzberg J. Development and validation of a rapid, aldehyde dehydrogenase bright-based cord blood potency assay. Blood. 2016 May 12;127(19):2346-54. doi: 10.1182/blood-2015-08-666990. Epub 2016 Mar 11. PMID 26968535
- [Result] Bakbak E, Krishnaraj A, Bhatt DL, Quan A, Park B, Bakbak AI, Bari B, Terenzi KA, Pan Y, Fry EJ, Terenzi DC, Puar P, Khan TS, Rotstein OD, Mazer CD, Leiter LA, Teoh H, Hess DA, Verma S. Icosapent ethyl modulates circulating vascular regenerative cell content: The IPE-PREVENTION CardioLink-14 trial. Med. 2024 Jul 12;5(7):718-734.e4. doi: 10.1016/j.medj.2024.03.009. Epub 2024 Mar 28. PMID 38552629